CLINICAL TRIAL: NCT05694533
Title: An Open Label, Fixed-sequence Study to Evaluate the Potential CYP3A4 Induction Effect of INDV-2000 Using Oral Midazolam as a Probe in Healthy Adults Participants
Brief Title: Study of Potential CYP3A4 Induction by INDV-2000 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INDV-2000-104; UG3DA050308 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INDV-2000 BID + Midazolam (Experimental): Participants will receive a single oral dose of 5 mg midazolam on Day 1. Participants will receive a dose of INDV-2000 twice a day (BID) from Days 2 to 15. On Day 15 participants will also receive a single oral dose of 5 mg midazolam co-administered with the INDV-2000 morning dose.
  Interventions: Drug: INDV-2000; Drug: Midazolam

INTERVENTIONS:
Drug: INDV-2000 — Capsules administered orally twice a day
  Other Names: C4X_3256
Drug: Midazolam — Midazolam syrup administered orally on Days 1 and 15

SUMMARY:
The purpose of this study is to investigate the potential for cytochrome P450 (CYP) 3A4 induction after dosing with INDV-2000 via use of midazolam as a probe.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
2. Body weight of a minimum of 50.0 kg at the screening visit and body mass index within the range 18.0 - 32.0 kg/m^2 (inclusive).
3. Male or female who is healthy as determined by medical evaluation.
4. Females will be of non-childbearing potential. Females of non-childbearing potential are considered women who:

   * Do not have a uterus, or
   * Are surgically sterile (eg, has undergone complete hysterectomy, bilateral oophorectomy, hysteroscopic sterilization, or tubal ligation), or
   * Have permanent cessation of ovarian function due to ovarian failure or surgical removal of the ovaries, or
   * Are post-menopausal as defined by 12 months or more of spontaneous amenorrhea as confirmed by a follicle-stimulating hormone (FSH) > 30 mIU/mL
5. Male participants agree to follow contraception guidelines specified in the Protocol.
6. Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting.
7. Capable of giving signed informed consent.

Exclusion Criteria:

1. Have an ongoing medical history of clinically significant neurological, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal (GI) disease, psychiatric or other disorder as judged by an Investigator that could potentially affect the study outcomes or compromise participant safety.
2. Have clinically significant abnormal biochemistry, hematology or urinalysis results as judged by an Investigator.
3. Have a history of narcolepsy or sleep apnea.
4. Have disorders that may interfere with drug absorption, distribution, metabolism and excretion processes.
5. Current active hepatic or biliary disease.
6. Participants with cholecystectomy < 90 days prior to screening.
7. Positive test results for human immunodeficiency virus (HIV)-1/HIV-2 antibodies, Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies.
8. Have a blood pressure reading outside of the following range: Systolic < 86 or > 149 mmHg; Diastolic < 50 or > 94 mmHg
9. Serious cardiac illness or other medical condition including, but not limited to:

   * Uncontrolled arrhythmias
   * History of congestive heart failure
   * QTcF > 450 msec for males and > 470 msec for females or history of prolonged QT syndrome
   * Myocardial infarction
   * Uncontrolled symptomatic angina
10. History of suicidal ideation within 30 days prior to providing written informed consent as evidenced by answering "yes' to questions 4 or 5 on the suicidal ideation portion of the C-SSRS completed at the screening visit or history of a suicide attempt (per the C-SSRS) in the 6 months prior to informed consent.
11. Healthy participants who are taking, or have taken, any prescribed or over-the-counter drugs (other than 2 grams of acetaminophen per 24-hour period as of Day 1, hormone replacement therapy, or thyroid hormone replacement therapy) or herbal remedies in the 14 days or 5 half-lives (whichever is longer) prior to first dose of study drug.
12. Treatment with any known drugs that are moderate or strong inhibitors/inducers of CYP3A4 or CYP2C19, including St. John's Wort, within 30 days prior to first dose of study drug.
13. Any consumption of food or drink containing poppy seeds, grapefruit or Seville oranges within 14 days prior to the first dose of study drug.
14. Regular alcohol consumption in males > 21 units per week and females > 14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
15. Positive test result for alcohol and/or drugs of abuse at screening or at check-in.
16. Female participant with a positive pregnancy test at the screening visit or at first check-in or who are lactating.
17. Concurrent treatment or treatment with an investigational drug or device within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
18. Blood donation of approximately 500 mL or more within 56 days or plasma donation within 7 days of screening.
19. Known hypersensitivity to INDV-2000 or any other ingredient in the INDV-2000 formulation.
20. Known hypersensitivity to midazolam or any other ingredient in midazolam HCl syrup.
21. Site staff and/or participants who have a financial interest in, or an immediate family member of either the site staff and/or Indivior employees, directly involved in the study.
22. Major surgical procedure (as defined by the Investigator) within 90 days prior to the first dose of study drug or still recovering from prior surgery.
23. Concurrent enrollment in another clinical study, unless it is an observational study.
24. Participants who are unable, in the opinion of the Investigator, to comply fully with the study requirements.
25. Any condition that, in the opinion of the Investigator or Indivior, would interfere with evaluation of the study drug or interpretation of participant safety or study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- INDV-2000 BID + Midazolam: Participants received a single oral dose of 5 mg midazolam on Day 1. Participants received a dose of INDV-2000 twice a day (BID) from Days 2 to 15. On Day 15 participants also received a single oral dose of 5 mg midazolam co-administered with the INDV-2000 morning dose.
  INDV-2000: Capsules administered orally twice a day
  Midazolam: Midazolam syrup administered orally on Days 1 and 15
Period: Overall Study
Arm/Group | INDV-2000 BID + Midazolam
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INDV-2000 BID + Midazolam
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Midazolam and 1-hydroxymidazolam
Time Frame: Day 1 and Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INDV-2000 BID + Midazolam
Number analyzed (Participants) | 20
ng/mL
  Midazolam Day 1 | 22.0 (47.2)
  Midazolam Day 15 | 18.5 (30.8)
  1-Hydroxymidazolam Day 1 | 9.92 (47.1)
  1-Hydroxymidazolam Day 15 | 7.97 (40.9)
Statistical Analysis 1: Comparison: INDV-2000 BID + Midazolam; The comparison is between Midazolam on Day 15 and Midazolam on Day 1; Test type: Other — Descriptive only; A random effects model was used to calculate the confidence interval; Geometric Mean Ratio = 0.84, 90% CI 2-sided [0.76 to 0.92] — Day 15/Day 1
Statistical Analysis 2: Comparison: INDV-2000 BID + Midazolam; The comparison is between 1-hydroxymidazolam on Day 15 and 1-hydroxymidazolam on Day 1; Test type: Other — Descriptive only; A random effects model was used to calculate the confidence interval; Geometric Mean Ratio = 0.80, 90% CI 2-sided [0.69 to 0.93] — Day 15/Day 1

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Midazolam and 1-hydroxymidazolam
Time Frame: Day 1 and Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | INDV-2000 BID + Midazolam
Number analyzed (Participants) | 20
hour*ng/mL
  Midazolam Day 1 | 57.2 (46.1)
  Midazolam Day 15 | 48.5 (36.3)
  1-Hydroxymidazolam Day 1 | 25.2 (35.2)
  1-Hydroxymidazolam Day 15 | 20.3 (32.6)
Statistical Analysis 1: Comparison: INDV-2000 BID + Midazolam; The comparison is between Midazolam on Day 15 and Midazolam on Day 1; Test type: Other — Descriptive only; A random effects model was used to calculate the confidence interval; Geometric Mean Ratio = 0.85, 90% CI 2-sided [0.78 to 0.92] — Day 15/Day 1
Statistical Analysis 2: Comparison: INDV-2000 BID + Midazolam; The comparison is between 1-hydroxymidazolam on Day 15 and 1-hydroxymidazolam on Day 1; Test type: Other — Descriptive only; A random effects model was used to calculate the confidence interval; Geometric Mean Ratio = 0.81, 90% CI 2-sided [0.74 to 0.89] — Day 15/Day 1

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Midazolam and 1-hydroxymidazolam
Time Frame: Day 1 and Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | INDV-2000 BID + Midazolam
Number analyzed (Participants) | 20
hour*ng/mL
  Midazolam Day 1 | 55.5 (45.5)
  Midazolam Day 15 | 46.9 (35.6)
  1-Hydroxymidazolam Day 1 | 23.2 (43.4)
  1-Hydroxymidazolam Day 15 | 20.1 (33.0)
Statistical Analysis 1: Comparison: INDV-2000 BID + Midazolam; The comparison is between Midazolam on Day 15 and Midazolam on Day 1; Test type: Other — Descriptive only; A random effects model was used to calculate the confidence interval; Geometric Mean Ratio = 0.85, 90% CI 2-sided [0.78 to 0.91] — Day 15/Day 1
Statistical Analysis 2: Comparison: INDV-2000 BID + Midazolam; The comparison is between 1-hydroxymidazolam on Day 15 and 1-hydroxymidazolam on Day 1; Test type: Other — Descriptive only; A random effects model was used to calculate the confidence interval; Geometric Mean Ratio = 0.87, 90% CI 2-sided [0.78 to 0.97] — Day 15/Day 1

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs will be defined as adverse events that start on or after the first dose of study drug.
Time Frame: From first dose of study drug to Day 22
Measure: Count of Participants; unit: Participants
Groups:
- Midazolam: Midazolam alone
- INDV-2000: INDV-2000 alone
- Midazolam + INDV-2000: INDV-2000 co-administered with midazolam
Arm/Group | Midazolam | INDV-2000 | Midazolam + INDV-2000
Number analyzed (Participants) | 20 | 20 | 20
Participants | 7 | 12 | 3

ADVERSE EVENTS:
Time Frame: 22 days
Description: All AEs and SAEs were collected from informed consent form signature until the end of study (EOS) Visit on Day 22 (±2 days) or at early termination. Any ongoing AEs at the time of the EOS Visit (ie, Day 22 [±2 days]) or at early termination were appropriately followed-up until resolution or 14 days after the EOS Visit or early termination.
Arm/Group | Midazolam | INDV-2000 | Midazolam + INDV-2000
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 12/20 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam (N=20) | INDV-2000 (N=20) | Midazolam + INDV-2000 (N=20)
SOMNOLENCE (Nervous system disorders) | 4 | 4 | 1
HEADACHE (Nervous system disorders) | 1 | 4 | 2
DIZZINESS (Nervous system disorders) | 2 | 1 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 3 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
FATIGUE (General disorders) | 2 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 2 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT05694533/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT05694533/SAP_001.pdf